CLINICAL TRIAL: NCT06202703
Title: Optimisation of Lymph Node Fine Needle Aspiration to Study Pneumococcal Vaccine-induced Immunity
Brief Title: Fine Needle aSpiration of Lymph nodEs to Study vAccine-induced Immunity
Acronym: SEA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Anna HE Roukens, Principal Investigator, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: U1111-1285-0005
Record Dates: First submitted 2023-05-23; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Vaccine-Preventable Diseases
MeSH Terms: conditions — Vaccine-Preventable Diseases | interventions — Pneumococcal Vaccines; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pneumococcal vaccination arm (Experimental): the participants will receive a registered pneumococcal vaccine according to manufacturers instructions
  Interventions: Drug: Pneumococcal Vaccine

INTERVENTIONS:
Drug: Pneumococcal Vaccine — vaccination with pneumococcal vaccine (PCV13)
  Other Names: vaccine with pneumococcal polysaccharides of 13 different serotypes conjugated to a protein (Prevnar13)

SUMMARY:
Rationale Causing a wide range of infectious diseases, including pneumonia, otitis media and meningitis, S. pneumoniae represents an important global health problem. Pneumococcal vaccines are clinically effective in preventing invasive pneumococcal disease, but the underlying immune response is likely to differ due to the inclusion of T cell epitopes in the conjugate, but not purified polysaccharide vaccine. However, these differences remain scantly studied. Lymph node fine needle aspiration (FNA) has been recently described to study vaccine-induced germinal centre responses in depth and represents a promising tool to study the underlying immune mechanisms of pneumococcal vaccines. Insight into the underlying immune mechanisms of vaccines could improve future vaccine design, e.g. by refining dosing intervals.

Objective Determine timing of peak germinal centre B cell frequency following pneumococcal vaccination.

Main trial endpoints The main trial endpoint is represented by the frequency of germinal centre B cells (BGC) in lymph node aspirates at various time points after vaccination, as measured by spectral flow cytometry. Both total BGC cells and S. pneumoniae polysaccharide-specific BGC frequencies will be determined.

Trial design Pilot intervention study without a comparator.

Trial population Healthy individuals between the age of 20 - 40

Interventions Subjects will be vaccinated once with Prevenar13. FNA of the draining lymph node will be performed and blood will be drawn at baseline, followed by weekly collection during the first four weeks, every other week between weeks 4 - 8 and a final collection time point after 12 weeks, resulting in a total of 8 sampling time points over the course of three months. Draining lymph node size will be assessed by ultrasound every other day during the first two weeks and then alongside lymph node FNA for the remainder of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants between the ages of 20 and 40 years old
* Participants should be generally healthy and without substantial co-morbidities, including all auto-immune diseases that are being actively treated with immunosuppressive therapy. Patients with chronic diseases that do not require immunosuppressive therapy and are stable, defined as not requiring change of therapy or hospitalization in the six weeks preceding study enrollment, might be eligible for this study.

Exclusion Criteria:

* BMI > 30 kg/m2
* Pregnancy at time of inclusion
* Breastfeeding during the course of the study
* Documented pneumococcal vaccination and/or infection
* Pneumococcal infection is defined as any infection that is microbiologically confirmed to be caused by S. pneumoniae (e.g. positive blood or sputum cultures for S. pneumoniae, positive urine S. pneumoniae antigen test)
* Documented HIV infection
* Documented primary immune disorder or primary coagulopathy
* Use of immunosuppressive medication or anticoagulants
* Known hypersensitivity to any of the vaccine components
* Recent (i.e. <4 weeks before inclusion) surgery in axillar area or major surgery elsewhere
* Vaccination with any vaccine < 1 month before inclusion
* Subjects vaccinated 1 - 6 months before enrolment can be included into the study. Study vaccine will be injected in the contralateral arm.
* Fever at time of inclusion

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
peak germinal center B cell count | 3 months
  frequency of germinal centre B cells (BGC) in lymph node aspirates will be measured at various time points after vaccination, as measured by spectral flow cytometry. Lymph node sampling will take place every week for the first 4 weeks, than every other week until week 8. Characterization of the lymphocytes in the lymph node aspirate will be performed by flow cytometry

SECONDARY OUTCOMES:
immune analysis of lymph node aspirates after pneumococcal vaccination | 3 months
  In addition to evaluating the frequency of (antigen-specific) BGC cells (outcome 1), we will perform phenotyping of these cells. Phenotyping includes measurement of activation markers, immunoglobulin class switching and markers associated with B cell differentiation.

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No
we will share data under restricted access, this is out institution's policy